CLINICAL TRIAL: NCT03057535
Title: Effect of Induced Metabolic Alkalosis by Sodium Bicarbonate Administration on the Ventilatory Response to Exercise in Healthy Adults
Brief Title: Impact of NaHCO3- on Exercise Hyperpnea
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Dennis Jensen, Ph.D., Assistant Professor, McGill University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A02-M19-15B
Record Dates: First submitted 2017-02-10; First posted 2017-02-20 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Pulmonary Ventilation
Keywords: Exercise; Sodium Bicarbonate; Ventilatory equivalent for carbon dioxide
MeSH Terms: conditions — Motor Activity | interventions — Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Bicarbonate (Experimental): Ingestion of sodium bicarbonate (0.3 g/kg of body mass)
  Interventions: Drug: Sodium Bicarbonate
- Sodium Chloride (Placebo Comparator): Ingestion of sodium chloride (4 g)
  Interventions: Drug: Sodium Chloride

INTERVENTIONS:
Drug: Sodium Bicarbonate
  Arms: Sodium Bicarbonate
Drug: Sodium Chloride
  Arms: Sodium Chloride

SUMMARY:
An abnormally high V̇E/V̇CO2 response to exercise is a key pathophysiological feature of patients with chronic cardiopulmonary disease that is associated with adverse health outcomes. It follows that any intervention capable of decreasing the V̇E/V̇CO2 response to exercise has the potential to improve clinical and/or patient-reported outcomes. The investigators of this trial will compare the effects of orally administered sodium chloride (4 g, placebo) and sodium bicarbonate (0.3 g/kg of body mass) on ventilation, breathing pattern, dynamic operating lung volume, gas exhange, cardiovascular, metabolic and symptom parameters during symptom-limited, high-intensity, constant-work-rate cycle exercise testing in healthy adults aged 20-40 years.

DETAILED DESCRIPTION:
The ventilatory response (V̇E) to exercise-induced increases in the rate of CO2 production (V̇CO2) depends on the regulated level of arterial PCO2 (PaCO2) and the dead space to tidal volume ratio (VD/VT).

An abnormally high V̇E/V̇CO2 response to exercise, reflecting a high VD/VT and/or low PaCO2 equilibrium point, is a key pathophysiological feature of patients with chronic cardiopulmonary disease, including heart failure, pulmonary arterial hypertension, interstitial lung disease and chronic obstructive pulmonary disease. In these patient groups, exercise ventilatory inefficiency is associated with: disease severity and progression; exercise intolerance; exertional breathlessness; and increased risk of hospitalization, major cardiac events and mortality. It follows that any intervention capable of decreasing the V̇E/V̇CO2 response to exercise has the potential to improve clinical and/or patient-reported outcomes. Unfortunately, our ability to enhance exercise ventilatory efficiency is limited by the fact that, with the possible exception of lung volume reduction surgery in chronic obstructive pulmonary disease and pulmonary vasodilator therapy in pulmonary arterial hypertension and heart failure, ventilation-perfusion abnormalities reflecting a high VD/VT are often irreversible.

A largely unexplored approach to decreasing the V̇E/V̇CO2 response to exercise is increasing the PaCO2 equilibrium point by inducing a metabolic alkalosis via administration of an alkalizing agent such as sodium bicarbonate (NaHCO3). Thus, the primary objective of this randomized, double blind, placebo controlled, crossover study was to test the hypothesis that increasing the PaCO2 equilibrium point via induced acute metabolic alkalosis by single-dose oral administration of NaHCO3 would decrease in the V̇E/V̇CO2 ratio at its lowest point ("nadir") during high-intensity constant-load cycle exercise testing in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smoking
* Habitually active
* Non-obese (Body Mass Index <30 kg/m2)
* Normal lung function on spirometry

Exclusion Criteria:

* Self-reported gastrointestinal, cardiovascular, vascular, respiratory, kidney, liver, musculoskeletal, endocrine, neuromuscular and/or metabolic disease/dysfunction
* Taking doctor prescribed medications other than oral contraceptives

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Ventilatory equivalent to carbon dioxide (V̇E/V̇CO2) at its lowest point ("nadir") during exercise | Participants will be followed until all study visits are complete, an expected average of 3 weeks
  The V̇E/V̇CO2 nadir will be identified as the lowest 30-sec average data point during constant-load cycle exercise testing

SECONDARY OUTCOMES:
Partial pressure of carbon dioxide in the arterialized capillary blood (PacCO2) | Time Frame: Participants will be followed until all study visits are complete, an expected average of 3 weeks
  PacCO2 (mmHg) will be measured at rest 90-min post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Jensen, Ph.D., Principal Investigator — McGill University
Locations (1):
- McGill University, Department of Kinesiology & Physical Education, Clinical Exercise & Respiratory Physiology Laboratory, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Exercise & Respiratory Physiology Laboratory (CERPL) of McGill University — http://www.mcgill.ca/cerpl